CLINICAL TRIAL: NCT06635902
Title: A Phase 2 Randomized Double-blind, Placebo-controlled Clinical Trial of Intravenous Citrulline for Vaso-occlusive Pain Episode in Hospitalized Patients With Sickle Cell Disease (CONQUER SCD Pain Trial)
Brief Title: Intravenous L-Citrulline for Vaso-occlusive Pain Episode in Sickle Cell Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Suvankar Majumdar (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Suvankar Majumdar, Chief of Hematology, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00000880; 1R61HL167806 (NIH)
Record Dates: First submitted 2024-10-07; First posted 2024-10-10 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Sickle Cell Disease; Vaso-occlusive Pain Episode
Keywords: sickle cell disease; sickle cell pain crisis; citrulline
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Citrulline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low dose intravenous L-citrulline (Experimental)
  Interventions: Drug: L-citrulline
- High dose intravenous L-citrulline (Experimental)
  Interventions: Drug: L-citrulline
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: L-citrulline — Intravenous L-citrulline (50 mg/kg + 9mg/kg/hr.) for 16 hours
  Arms: High dose intravenous L-citrulline
Other: Placebo — Isotonic normal saline
  Arms: Placebo
Drug: L-citrulline — Intravenous L-citrulline (25 mg/kg + 9mg/kg/hr.) for 16 hours
  Arms: Low dose intravenous L-citrulline

SUMMARY:
The goal of this clinical trial is to learn if intravenous citrulline works to treat acute pain in hospitalized patients with sickle cell disease. It will also learn about the safety of intravenous citrulline. The main questions it aims to answer are:

* Does intravenous citrulline decrease the duration of sickle cell pain during hospitalization
* What medical problems do participants have when taking intravenous citrulline? Researchers will compare intravenous citrulline to a placebo (a look-alike substance that contains no drug) to see if intravenous citrulline works to treat acute pain.

Participants will:

* Receive baseline tests and intravenous citrulline for 16 hours during the hospital stay
* After hospital discharge, visit the clinic in about 30 days for checkup and tests

DETAILED DESCRIPTION:
This is a single-center phase 2 randomized double-blind, placebo-controlled trial of intravenous L-citrulline for sickle cell patients ages 4 to 21 years experiencing a vaso-occlusive pain crisis episode (VOE). Eligible subjects will have a documented history of sickle cell disease and inpatient hospitalization for treatment of acute pain with parenteral opioid. Subjects will be randomized to receive high dose intravenous L-citrulline, low dose intravenous L-citrulline or placebo in addition to standard of care. Subjects will be followed closely to evaluate time-to-crisis resolution as the primary outcome defined by time from first dose of intravenous study drug/placebo to the last dose of parenteral opioid prior to hospital discharge. Participants will be monitored for any adverse events including 30-day re-hospitalization rates. Total opioid consumption during the time-to-crisis resolution will be compared between the three arms. In addition, exploratory outcomes will be evaluated for pain score, tissue blood flow, genetic and candidate biomarkers related to vaso-occlusion.

Objectives Primary Objective

• To demonstrate the efficacy of intravenous L-citrulline in reducing the time-to-crisis resolution in sickle cell subjects experiencing a vaso-occlusive pain crisis episode (VOE).

Secondary Objectives

* To evaluate the safety of intravenous L-citrulline in the treatment of VOE
* To determine if intravenous L-citrulline improves cumulative opioid consumption during the treatment of VOE Exploratory Objectives
* To determine if intravenous L-citrulline improves pain scores during the hospitalization
* To determine if intravenous L-citrulline improves 30-day re-hospitalization rates
* To determine the pharmacokinetic (PK) profile of intravenous L-citrulline
* To evaluate whether intravenous L-citrulline improves tissue blood flow and candidate biomarkers related to vaso-occlusion.
* To assess whether genetic single nucleotide polymorphisms related to the nitric oxide pathway influence study outcomes

ELIGIBILITY:
Inclusion Criteria:

* Sickle cell disease (all genotypes)
* Patients with sickle cell disease ages 4 to 21 years old
* Presence of sickle cell vaso-occlusive pain episode requiring hospitalization and parenteral opioid therapy
* Able to randomize to study drug/placebo within 12 hours of first dose of parenteral opioid in the Emergency Department

Exclusion Criteria:

* Current pain lasting >3 days.
* >9 hospitalizations in the prior year
* Presence of any other complication related to sickle cell disease requiring the hospitalization such as splenic sequestration, hepatic sequestration, stroke, transient ischemic attack, etc.
* History of opioid use disorder, chronic pain or medical regimen requiring daily opioid use.
* Severe anemia (hemoglobin <6g/dL)
* Pregnant (as confirmed by a positive urine pregnancy test) or lactating female.
* Alanine/aspartate transferase >2x upper limit of normal laboratory range for age.
* Subject has the following serum creatinine:

  * Age 4 to 13 years > 0.9 mg/dL
  * Age 14 to 17 years 1.0 mg/dL
  * Age ≥18 years >1.5mg/dL
* Presence of acute chest syndrome, sepsis, bacterial infection, hemodynamic instability
* Use of L-glutamine
* History of allergic reaction to L-citrulline products

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 99 (Estimated)
Dates: Start 2024-12-22 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Time-to-crisis resolution | Baseline to 30 days
  Change in time-to-crisis resolution as defined by the time (in hours) from first dose of intravenous study drug or placebo to the time of last dose of intravenous opioid during hospitalization

SECONDARY OUTCOMES:
Safety | Baseline to 30 days
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0
Opioid consumption | Baseline to 30 days
  Change in cumulative opioid consumption (calculated in morphine equivalents) from time of study drug administration to last dose of IV/oral opioid during hospitalization
Pain scores | Baseline to 30 days
  Change in baseline pain scores will be recorded from a 0-10 scale, 10 is worst pain

OTHER OUTCOMES:
Citrulline and arginine bioavailability | Baseline to 30 days
  Change in baseline citrulline and arginine concentration during hospitalization and 30 day follow up/
Nitric oxide | Baseline to 30 days
  Change in baseline nitric oxide concentration during hospitalization and 30 day follow up
Cytokine interleukin IL-1ß | Baseline to 30 days
  Change in baseline plasmatic levels of IL-1ß concentration during hospitalization and 30 day follow up
Mitochondrial function | Baseline to 30 days
  Mitochondrial respiratory complex activities will be measured to estimate mitochondrial function. Change in baseline mitochondrial respiratory complex activity during hospitalization and 30 day follow up
Genetic | Baseline
  DNA to test specific genetic polymorphisms related to nitric oxide pathway

CONTACTS AND LOCATIONS:
Overall Officials: Suvankar Majumdar, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be shared
Supporting Information: ICF
Time Frame: Beginning 3 months and ending 3 years after the publication of results
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP). For more information or to submit a request, please contact smajumdar@childrensnational.org